CLINICAL TRIAL: NCT00002373
Title: A Phase I/II Trial to Evaluate the Tolerability, Anti-CMV Activity and Pharmacokinetics of 1263W94 Following Multiple Oral Administration of Escalating Doses in HIV-Infected Patients With Asymptomatic CMV Shedding
Brief Title: The Safety and Effectiveness of Different Dose Levels of 1263W94 in the Treatment of Cytomegalovirus (CMV) of the Eyes in HIV-Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 263A; CMAA1003
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-11

CONDITIONS: Cytomegalovirus Infections; HIV Infections
Keywords: Cytomegalovirus; Cytomegalovirus Infections; Administration, Oral; Acquired Immunodeficiency Syndrome; Antiviral Agents; Virus Shedding; Viral Load
MeSH Terms: conditions — Cytomegalovirus Infections; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — maribavir

INTERVENTIONS:
Drug: Maribavir

SUMMARY:
To evaluate the safety and tolerability of multiple escalating doses of 1263W94 administered orally for 28 days in HIV infected patients with asymptomatic CMV shedding. To obtain preliminary evidence of the in vivo anti CMV activity of different doses of 1263W94 in humans based on quantitative reduction of CMV load in semen and if possible in other biological fluids and to explore the dose response relationship in the anti-CMV activity of 1263W94.

DETAILED DESCRIPTION:
HIV seropositive men stratified based on CMV titer in semen at the Pre-Screen visit (30 days prior to entry). Patients with a CMV titer >= 5000 PFU/ml and a positive result upon qualitative urine CMV culture may be eligible for entry into the main group and patients with a CMV titer < 5000 PFU/ml may be eligible for entry into the satellite group. Patients will on 1263W94 for 4 weeks. Patients will be present for clinic visits on study days 1, 7, 14, 21, and 28. They will return to the clinic for post treatment evaluations on study days 42 and 56.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

Stable, chronically administered concomitant therapy for HIV infection and opportunistic diseases if patient has been on the regimen for at least one month prior to study entry.

Patients must have:

Required of Main group:

* Minimum CMV titer of 5000 PFU/ml in semen by quantitative CMV culture on one occasion within 30 days of entry.
* Demonstrating positive result of qualitative CMV culture in urine on one occasion within 30 days of entry.

Required of Satellite group:

* Must have CD4+ < 150 c/mm3 (or 10% of total lymphocytes) at screen.

Required of both groups:

* HIV infection.
* Life expectancy > 6 months.
* Able to comply with protocol requirements/instructions and likely to complete all study visits and evaluations as planned.

Prior Medication:

Allowed:

Stable, chronically administered concomitant therapy for HIV infection and opportunistic diseases for at least one month prior.

Exclusion Criteria

Co-existing Condition:

Patients with any of the following symptoms or conditions are excluded:

* Active CMV disease (retinitis, colitis, encephalitis, pneumonitis, etc.).
* Visual symptoms or signs suggestive of CMV disease (e.g., floaters, visual field defects, decreased visual acuity); Unless CMV disease is excluded via ophthalmoscopy examination.
* Active hepatitis, obstructive hepatobiliary diseases or cirrhosis.
* Gastrointestinal disorders which, in the judgement of the investigator, might interfere with oral dosing and drug absorption or may be indicative of CMV disease e.g., chronic nausea or vomiting, active bowel disease or persistent diarrhea.
* Diagnosis of chronic diseases such as diabetes or hypoglycemia, epilepsy, ongoing Grade II peripheral neuropathy, congestive heart failure, cardiomyopathy, other organ dysfunctions, etc., which in the opinion of the investigator, would compromise the safety or compliance of the patient.
* Participation in other investigational trials.
* Patients who are so debilitated as a result of their HIV disease or associated illness or therapies such that, in the investigator's opinion, the condition may interfere with the study assessments or the patient's ability to complete the entire study per protocol requirements.

Concurrent Medication:

Excluded:

Systemic therapy for visceral malignancy.

Concurrent Treatment:

Excluded:

Treatment with radiation therapy for visceral malignancy.

Patients with any of the following prior symptoms or conditions are excluded:

* History of CMV disease (such as retinitis, colitis, encephalitis, pneumonitis, etc.)
* Known history of lactose intolerance.

Prior Medication:

Excluded:

* Systemic therapy for visceral malignancy within 2 months prior to entry.
* Prior treatment with ganciclovir, foscarnet, cidofovir, or other investigational anti-CMV drugs (e.g., intravenous acyclovir, lobucavir, valacyclovir) within 2 months prior to entry.
* Treated with interferons, immunomodulators or CMV hyperimmune globulin within 1 month prior to entry.
* Any investigational therapies within 1 month prior of study entry.

Prior Treatment:

Excluded:

* Treatment with radiation therapy for visceral malignancy within 2 months prior to entry.
* Treatment with any investigational treatments within 1 month of study entry.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Univ of California/ San Francisco / Dept of Medicine, San Francisco, California
  - Dr Jacob Lalezari, San Francisco, California